CLINICAL TRIAL: NCT03873194
Title: Use of Meditation as a Complementary Therapy in the Treatment of Gestational Hypertension
Brief Title: Meditation as Complementary Treatment for Chronic Hypertension in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 93028218.7.0000.0068
Record Dates: First submitted 2019-02-27; First posted 2019-03-13 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2020-11

CONDITIONS: Hypertension, Pregnancy-Induced; Hypertension in Pregnancy; Hypertension
Keywords: systemic arterial hypertension; hypertension; hypertension, pregnancy-induced; pre-eclampsia; meditation; randomized clinical Trial
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension; Pre-Eclampsia | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: The objective of this study is assess the effect of meditation as a complementary therapy in hypertensive pregnant women.
  The method used will be a randomized, controlled and blinded clinical trial, where meditation is going to be offered between March 2019 and July 2020 at the Obstetrics Clinic of Hospital of Clinics, Faculty of Medicine, University of São Paulo. Patients are going to be randomly assigned to two groups: Group I, patients who are going to practice meditation and Group II, patients that will receive only the usual outpatient care.
  The allocation will be performed according to CONSORT criteria and sequential within two classifications of diastolic blood pressure values.
  Differences between the means of the variables (blood pressure levels and questionnaires about life quality, anxiety, resilience and mindfulness) will be compared between the groups. Values of p<0,05 will be considered significant.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Blinding will be used in the following manner: after informed consent, an auxiliary researcher will randomly allocate participants to 2 research groups (Group A or Group B). After this step, the auxiliary researcher will collect data for the study and will refer the patient for the usual treatment or for the usual treatment and also meditation.
  The lead researcher will not have access to the data that was collected at the beginning of the study by the auxiliary researcher before the end of the intervention step. He will analyse the results without knowing which patients were in which group (A or B). Only after statistical analysis the groups composition will be revealed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation group (Experimental): Patients who are going to practice meditation and will receive only the usual outpatient care, with the aim of observing reduction of systemic blood pressure in this period.
  Interventions: Other: Meditation; Other: conventional treatment
- conventional treatment (Other): Patients that will receive only the usual outpatient care, with the aim of observing the systemic blood pressure in this period.
  Interventions: Other: conventional treatment

INTERVENTIONS:
Other: Meditation — Participants will be instructed to find a comfortable position, with a straight back, feeling the general state of their bodies (tensions, pains, heat, cold, etc.), to relax and pay attention to their own breathing, being aware of the air that gets into and out of the lungs. The women will be told that whenever their attention disperses (to another focus such as a thought, a sound, a body sensation, a judgment, etc.) they should go back to the original focus (breathing) with no feeling/judgment about the loss of focus. The practice involves focus and attention exercises and the gradual insertion of other anchors (focus points) as participants improve their skills in this practice.
  Arms: Meditation group
Other: conventional treatment — Early prenatal care, when possible, is recommended as the first measure. Prenatal appointments usually take place fortnightly or weekly for hypertensive pregnant women. Extensive lab testing including specific tests for the first trimester, as well as tests for the diagnosis of superimposed pre-eclampsia and for the evaluation of lesions in target organs.
  Drug treatment is only used when non-drug measures against hypertension are inefficient to decrease blood pressure levels and diastolic pressure is 90 mmHg or higher (in the first half of pregnancy) and over 100 mmHg (after 20 weeks).

SUMMARY:
Pregnancy relates to arterial hypertension; it is an aggravating factor for pre-existing chronic arterial hypertension or a trigger for preeclampsia in normotensive women. The gestational hypertensive disease is managed conventionally with the pregnant woman's hospitalization and/or the use of antihypertensive medications. Nevertheless, this treatment may present some risks. The investigators seek to determine whether the intervention compared to the control can reduce the increase in blood pressure that pregnant women in the transition from the 2nd to the 3rd trimester.

DETAILED DESCRIPTION:
Primary research question:

Can meditation decrease the mean increase in diastolic blood pressure in pregnant hypertensive women at the transition from the second to the third trimester of gestation?

Secondary research question:

Can meditation decrease the mean increase in systolic blood pressure in pregnant hypertensive women at the transition from the second to the third trimester of gestation?

Does meditation practice increases (or decreases) the likelihood of change in Resilience indicators?

Does meditation practice increase (or decrease) the likelihood of change in anxiety and depression indicators?

Does meditation practice increase (or decrease) the likelihood of change in mindfulness indicators?

Does meditation practice increase (or decrease) the likelihood of change in quality of life indicators?

ELIGIBILITY:
Inclusion Criteria:

1. Pre-existing hypertension.
2. Single pregnancy, with gestational age between 20th and 24th weeks, with uncomplicated systemic arterial hypertension.
3. Prenatal follow-up in a high-risk pregnancy clinic.
4. No personal background of depression or psychiatric disorders.
5. No serious heart disease.
6. No illicit drugs and/or alcohol use.
7. Acceptance of the informed consent.
8. To follow the practice used in the study, the subjects are required to have an available phone in order to download an app which contains an audio guide for this purpose.

Exclusion Criteria:

1. Diagnosis of depression and psychiatric disorders during pregnancy.
2. Patients who do not return to follow-up or who want to quit the study.
3. To practice meditation.

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Comparison the means of diastolic blood pressure of pregnant women's between intervention group and control group. | 8 weeks
  Diastolic blood pressure control in pregnant women with chronic hypertension between intervention group (meditation practice) and control group, in the transition from the second to the third trimester of pregnancy, when there is a physiologic increase in arterial pressure.
  The diastolic pressure check will be in outpatient consultation with intervals of 15 days, during 8 weeks.
  The device used for checking the pressure will be the GAMMA XXL LF of Heine General Medicine.
  All blood pressure checks either in the intervention group or control group will be performed on the same device.
Comparison the means of systolic blood pressure of pregnant women's between intervention group and control group. | 8 weeks
  Systolic blood pressure control in pregnant women with chronic hypertension between intervention group (meditation practice) and control group, in the transition from the second to the third trimester of pregnancy, when there is a physiologic increase in arterial pressure.
  The systolic pressure check will be in outpatient consultation with intervals of 15 days, during.
  The device used for checking the pressure will be the GAMMA XXL LF of Heine General Medicine.
  All blood pressure checks either in the intervention group or control group will be performed on the same device.

SECONDARY OUTCOMES:
Assessment of quality of life with World Health Organization instrument for evaluating quality of life (Whoqol-bref) questionnaire. | 8 weeks
  Checking potential increases or decreases in the quality life indicator during pregnancy using the Whoqol-Bref questionnaire as a result measure.
  The questionnaire will be applied at the entrance of the participant in the study and at the end of the 8 weeks.
  This questionnaire is composed of four domains of quality of life, totaling 24 questions.
  The answers follow a Likert scale (from 1 to 5) and the domain scores for the WHOQOL-BREF were calculated by multiplying the mean of all items included within the domain by four. Potential scores for all domain scores, therefore, range from 4-20.
  Only the total quality of life score will be considered in this study. For this study, a larger score on the Whoqol-Bref demonstrates a better outcome for the group performing the meditation intervention.
Assessment of anxiety and depression with The Hospital Anxiety and Depression Scale (HADS). | 8 weeks
  Checking potential increase or decreases of anxiety and depression indicators during pregnancy using the HADS Scale as a result measure.
  The questionnaire will be applied at the entrance of the participant in the study and at the end of the 8 weeks.
  The Hospital Anxiety and Depression Scale (HADS) consist of 14 questions. It was divided into an Anxiety subscale (HADS-A) consist of 07 questions and a Depression subscale (HADS-D) consist of 07 questions both containing seven intermingled items.
  Each items can be scored from zero (0) to three (3), composing a maximum score of 21 points for each sub-scale.
  * HAD-anxiety: no anxiety from 0 to 8, with anxiety ≥ 9;
  * HAD-depression: without depression from 0 to 8, with depression ≥ 9.
  For this study, a larger score on the Resilience Scale demonstrates a worst outcome for the group performing the meditation intervention.
Assessment of the capacity to adapt and restore equilibrium to their lives and avoid the potentially deleterious effects of stress with Resilience Scale. | 8 weeks
  Checking potential increase or decreases of the capacity to adapt and restore equilibrium to their lives and avoid the potentially deleterious effects of stress, during pregnancy using the Resilience Scale as a result measure.
  The questionnaire will be applied at the entrance of the participant in the study and at the end of the 8 weeks.
  The Resilience Scale is the scale that consist of 25 questions concerning the capacity to adapt and restore equilibrium to their lives to be rated on a 7-point scale
  The Likert scale ranged from (1) disagree to (7) agree, with higher scores reflecting higher levels of trait mindfulness.
  Possible scores range from 25 to 175 with higher scores reflecting higher resilience.
  For this study, a larger score on the Resilience Scale demonstrates a better outcome for the group performing the meditation intervention.
Assessment on the presence or absence of attention to and awareness of what is occurring in the present, that differentiates meditation practitioners from others, with Mindful Attention Awareness Scale (MAAS) | 8 weeks
  Checking potential increase or decreases on the presence or absence of attention to and awareness of what is occurring in the present, that differentiates meditation practitioners from others, during pregnancy using the MAAS as a result measure.
  The questionnaire will be applied at the entrance of the participant in the study and at the end of the 8 weeks.
  The Mindful Attention Awareness Scale is the unidimensional scale that consists of 15 questions concerning attention or awareness in routine situations to be rated on a 6-point scale on how frequently or infrequently the teste experiences those situations.
  The Likert scale ranged from (1) almost always to (6) almost never, with higher scores reflecting higher levels of trait mindfulness.
  The lowest possible value to be achieved when answering this scale is 15 and the highest possible value is 90.
  For this study, a larger score on the MAAS scale demonstrates a better outcome for the group performing the meditation intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gow AJ, Bastin ME, Munoz Maniega S, Valdes Hernandez MC, Morris Z, Murray C, Royle NA, Starr JM, Deary IJ, Wardlaw JM. Neuroprotective lifestyles and the aging brain: activity, atrophy, and white matter integrity. Neurology. 2012 Oct 23;79(17):1802-8. doi: 10.1212/WNL.0b013e3182703fd2. PMID 23091073
- [Background] Himelstein S. Meditation research: the state of the art in correctional settings. Int J Offender Ther Comp Criminol. 2011 Jun;55(4):646-61. doi: 10.1177/0306624X10364485. Epub 2010 Mar 23. PMID 20332328
- [Background] Bernstein PS, Martin JN Jr, Barton JR, Shields LE, Druzin ML, Scavone BM, Frost J, Morton CH, Ruhl C, Slager J, Tsigas EZ, Jaffer S, Menard MK. Consensus Bundle on Severe Hypertension During Pregnancy and the Postpartum Period. J Obstet Gynecol Neonatal Nurs. 2017 Sep-Oct;46(5):776-787. doi: 10.1016/j.jogn.2017.05.003. Epub 2017 Jul 11. PMID 28709727
- [Background] Fitton CA, Steiner MFC, Aucott L, Pell JP, Mackay DF, Fleming M, McLay JS. In-utero exposure to antihypertensive medication and neonatal and child health outcomes: a systematic review. J Hypertens. 2017 Nov;35(11):2123-2137. doi: 10.1097/HJH.0000000000001456. PMID 28661961
- [Background] Ospina MB, Bond K, Karkhaneh M, Tjosvold L, Vandermeer B, Liang Y, Bialy L, Hooton N, Buscemi N, Dryden DM, Klassen TP. Meditation practices for health: state of the research. Evid Rep Technol Assess (Full Rep). 2007 Jun;(155):1-263. PMID 17764203
- [Background] Kozasa EH, Radvany J, Barreiros MA, Leite JR, Amaro E Jr. Preliminary functional magnetic resonance imaging Stroop task results before and after a Zen meditation retreat. Psychiatry Clin Neurosci. 2008 Jun;62(3):366. doi: 10.1111/j.1440-1819.2008.01809.x. No abstract available. PMID 18588603
- [Background] Stahl JE, Dossett ML, LaJoie AS, Denninger JW, Mehta DH, Goldman R, Fricchione GL, Benson H. Correction: Relaxation Response and Resiliency Training and Its Effect on Healthcare Resource Utilization. PLoS One. 2017 Feb 21;12(2):e0172874. doi: 10.1371/journal.pone.0172874. eCollection 2017. PMID 28222185
- [Background] Mulder EJ, Robles de Medina PG, Huizink AC, Van den Bergh BR, Buitelaar JK, Visser GH. Prenatal maternal stress: effects on pregnancy and the (unborn) child. Early Hum Dev. 2002 Dec;70(1-2):3-14. doi: 10.1016/s0378-3782(02)00075-0. PMID 12441200
- [Background] Vieten C, Astin J. Effects of a mindfulness-based intervention during pregnancy on prenatal stress and mood: results of a pilot study. Arch Womens Ment Health. 2008;11(1):67-74. doi: 10.1007/s00737-008-0214-3. Epub 2008 Mar 3. PMID 18317710
- [Background] Beddoe AE, Lee KA. Mind-body interventions during pregnancy. J Obstet Gynecol Neonatal Nurs. 2008 Mar-Apr;37(2):165-75. doi: 10.1111/j.1552-6909.2008.00218.x. PMID 18336440
- [Background] Beddoe AE, Paul Yang CP, Kennedy HP, Weiss SJ, Lee KA. The effects of mindfulness-based yoga during pregnancy on maternal psychological and physical distress. J Obstet Gynecol Neonatal Nurs. 2009 May-Jun;38(3):310-9. doi: 10.1111/j.1552-6909.2009.01023.x. PMID 19538619
- [Background] van den Heuvel MI, Donkers FC, Winkler I, Otte RA, Van den Bergh BR. Maternal mindfulness and anxiety during pregnancy affect infants' neural responses to sounds. Soc Cogn Affect Neurosci. 2015 Mar;10(3):453-60. doi: 10.1093/scan/nsu075. Epub 2014 Jun 12. PMID 24925904
- [Background] Narendran S, Nagarathna R, Narendran V, Gunasheela S, Nagendra HR. Efficacy of yoga on pregnancy outcome. J Altern Complement Med. 2005 Apr;11(2):237-44. doi: 10.1089/acm.2005.11.237. PMID 15865489
- [Background] Narendran S, Nagarathna R, Gunasheela S, Nagendra HR. Efficacy of yoga in pregnant women with abnormal Doppler study of umbilical and uterine arteries. J Indian Med Assoc. 2005 Jan;103(1):12-4, 16-7. PMID 16008324
- [Background] van den Heuvel MI, Johannes MA, Henrichs J, Van den Bergh BR. Maternal mindfulness during pregnancy and infant socio-emotional development and temperament: the mediating role of maternal anxiety. Early Hum Dev. 2015 Feb;91(2):103-8. doi: 10.1016/j.earlhumdev.2014.12.003. Epub 2015 Jan 8. PMID 25577496
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. Int J Surg. 2011;9(8):672-7. doi: 10.1016/j.ijsu.2011.09.004. Epub 2011 Oct 13. No abstract available. PMID 22019563
- [Background] Fossaluza V, Diniz JB, Pereira Bde B, Miguel EC, Pereira CA. Sequential allocation to balance prognostic factors in a psychiatric clinical trial. Clinics (Sao Paulo). 2009;64(6):511-8. doi: 10.1590/s1807-59322009000600005. PMID 19578654
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Wagnild GM, Young HM. Development and psychometric evaluation of the Resilience Scale. J Nurs Meas. 1993 Winter;1(2):165-78. PMID 7850498